CLINICAL TRIAL: NCT02677506
Title: A Randomized Comparison of Infraclavicular and Supraclavicular Brachial Plexus Blocks for Elbow Surgery
Brief Title: Infraclavicular or Supraclavicular Brachial Plexus Blocks for Elbow Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101723
Record Dates: First submitted 2016-01-12; First posted 2016-02-09 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Cubital Tunnel Syndrome; Biceps Tendon Rupture
Keywords: elbow
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supraclavicular (Experimental): Supraclavicular brachial plexus block will be done.
  Interventions: Procedure: Supraclavicular
- Infraclavicular (Active Comparator): Infraclavicular brachial plexus block block will be done.
  Interventions: Procedure: Infraclavicular

INTERVENTIONS:
Procedure: Supraclavicular — Brachial plexus block with supraclavicular approach
  Arms: Supraclavicular
Procedure: Infraclavicular — Brachial plexus block with infraclavicular approach
  Arms: Infraclavicular

SUMMARY:
This study compares the infraclavicular approach to supraclavicular approach of brachial plexus block for elbow surgery.

DETAILED DESCRIPTION:
Traditionally, infraclavicular as well as supraclavicular approaches to brachial plexus have been recommended for elbow surgery. Supraclavicular approach is considered to have a more rapid onset. However, investigators have noticed that the supraclavicular approach needs more supplementation if it is used for elbow surgery. Therefore more and more anesthesiologists now choose the infraclavicular approach for elbow surgery (though both approaches are recommended in the text books).

None of the published studies have addressed if one approach is indeed superior to the other specifically for elbow surgery. Therefore the investigators propose to undertake a study that will evaluate the two approaches to the brachial plexus specifically for elbow surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ambulatory elbow surgery under block
* ASA 1-3

Exclusion Criteria:

* Narcotic dependent
* Severe systemic illness
* Refusal of block
* localized infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time to completion of block | 30 minutes
  A clock will be used to assess this outcome. Complete sensory block in all dermatomes will be tested with ice.

SECONDARY OUTCOMES:
Readiness for surgery | 60 minutes
  A clock will be used to assess this outcome. Complete sensory and motor block at the time of incision will be considered readiness of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — Western University
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No